CLINICAL TRIAL: NCT03130842
Title: Comparing Efficacy of Oral Midazolam and Sublingual Alprazolam in Reducing Anxiety and Pain/Discomfort Related to Diagnostic Upper Gastrointestinal Endoscopy in Adults
Brief Title: Premedication With Alprazolam and Midazolam for Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Elham Tabesh, Dr., Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 395569
Record Dates: First submitted 2017-04-03; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Diagnostic Esophagogastroduodenoscopy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublingual alprazolam (Active Comparator)
  Interventions: Drug: Sublingual alprazolam
- Oral midazolam (Active Comparator)
  Interventions: Drug: Oral midazolam

INTERVENTIONS:
Drug: Sublingual alprazolam — Patients receive one dose of oral formulation of alprazolam 0.5 mg for sublingual-administered at least 30 minutes before the procedure.
  Arms: Sublingual alprazolam
Drug: Oral midazolam — Patients receive one dose of intravenous formulation of alprazolam 7.5 mg for oral-administered (in syrup with apple juice) at least 30 minutes before the procedure.
  Arms: Oral midazolam

SUMMARY:
Diagnostic upper GI endoscopy can be uncomfortable and stressful for many patients. Various methods are available for sedation during this procedure. Because of some side effects related to intravenous administration of sedatives, oral administration of these drugs is under attention. Alprazolam is a benzodiazepine which is used mainly in treatment of anxiety. Intravenous midazolam is being used by some centers for sedation during endoscopy, but the oral form can also be used with probably same efficacy. Hence, investigators compare the efficacy/safety of oral midazolam and sublingual alprazolam as for sedation during this procedure. Investigators hypothesize that sublingual alprazolam is as effective as oral midazolam in reducing anxiety and pain/discomfort related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Referring for upper GI endoscopy
* Age 18 to 65 years
* First experience of upper GI endoscopy
* Class I or II of American Anesthesiology Association
* Willingness to participate

Exclusion Criteria:

* Severe psychiatric, neurological, cardio-vascular, or renal disorders
* History of allergy or intolerance to benzodiazepines or lidocaine
* History of upper GI surgery
* Pregnancy or lactation
* GI anomalia during endoscopy
* Need for therapeutic procedures during endoscopy
* Active bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-09-17 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Discomfort assessed by patients on a 11-point numeric rating scales about 5 minutes after the procedure when patients are fully awake | 5 minutes after the procedure
  Procedure related discomfort is assessed by patients on a 11-point numeric rating scales about 5 minutes after the procedure when patients are fully awake.
Change in anxiety | At baseline and at 30 minutes after medication
  Procedure related anxiety is assessed by patients on a 11-point numeric rating scales at baseline and then at 30 minutes after the medication.

SECONDARY OUTCOMES:
Satisfaction is assessed by patients on a 11-point numeric rating scales about 5 minutes after the procedure when patients are fully awake. | 5 minutes after the procedure
  Procedure related satisfaction is assessed by patients on a 11-point numeric rating scales about 5 minutes after the procedure when patients are fully awake.
Tolerance is assessed by patients from no compliance (0) to excellent compliance (4) about 5 minutes after the procedure when patients are fully awake. | 5 minutes after the procedure
  Tolerance is assessed by patients from no compliance (0) to excellent compliance (4) about 5 minutes after the procedure when patients are fully awake.
Duration of the procedure | From endoscope insertion to endoscope removal
  Duration of the procedure is defined as time (minute) from endoscope insertion to endoscope removal.
Hypotension | At baseline, 30 minutes after medication, at the beginning of procedure, and then every 5 minutes for 30 minutes.
  Blood pressure is monitored from baseline to 30 minutes after beginning of the procedure, with 5 minutes intervals. Hypotension episode is defined as systolic blood pressure of < 90 mm Hg
Bradycardia | At baseline, 30 minutes after medication, at the beginning of procedure, and then every 5 minutes for 30 minutes.
  Heart rate is monitored from baseline to 30 minutes after beginning of the procedure, with 5 minutes intervals. Bradycardia episode is defined as heart rate of < 60 bpm.
Desaturation | At baseline, 30 minutes after medication, at the beginning of procedure, and then every 5 minutes for 30 minutes.
  Arterial O2 saturation is monitored from baseline to 30 minutes after beginning of the procedure, with 5 minutes intervals. Desaturation episode is defined as as arterial oxygen saturation of < 90%.

CONTACTS AND LOCATIONS:
Overall Officials: Vahid Sebghatolahi, MD, Study Director — Isfahan University of Medical Sciences
Locations (1):
- Department of Gastroenterology, Alzahra Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available based on the IUMS policy

REFERENCES:
- [Background] Shavakhi A, Soleiman S, Gholamrezaei A, Khodadoostan M, Shavakhi S, Tahery A, Minakari M. Premedication with sublingual or oral alprazolam in adults undergoing diagnostic upper gastrointestinal endoscopy. Endoscopy. 2014 Aug;46(8):633-9. doi: 10.1055/s-0034-1377305. Epub 2014 Jun 30. PMID 24977401